CLINICAL TRIAL: NCT00002048
Title: The Efficacy and Safety of Retrovir in Patients Infected With HIV Who Are Asymptomatic (CDC Group II) or Have Persistent Generalized Lymphadenopathy (CDC Group III)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 014J; 21
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1989-09

CONDITIONS: Lymphatic Disease; HIV Infections
Keywords: Acquired Immunodeficiency Syndrome; Zidovudine
MeSH Terms: conditions — Lymphatic Diseases; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Zidovudine

INTERVENTIONS:
Drug: Zidovudine

SUMMARY:
To evaluate the safety and tolerance of chronic administration of Retrovir (AZT) in HIV-infected adult patients without clinical manifestations of disease. To assess the efficacy of AZT therapy in the treatment of HIV disease in these patients.

ELIGIBILITY:
Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* Prior history of a malignancy other than cutaneous basal cell or cervical carcinomas.
* Other significant, chronic underlying medical illness which would impair study completion.
* Liver dysfunction as demonstrated by lab results.
* Laboratory evidence of compromised bone marrow function.

Concurrent Medication:

Excluded:

* Any other experimental agents.
* Any probenecid-containing product.

Patients are excluded if they have a history of symptoms characteristic of CDC class I or IV including any of the following:

* Unintentional weight loss of greater than 10 lbs, or more than 10 percent of usual body weight within the last 16 weeks.
* Unexplained fever > 38.5 degrees C on more than 14 consecutive days or on more than 15 days in the previous 30-day period.
* Unexplained diarrhea defined by = or > 2 liquid stools per day persisting for = or > 14 days or 15 days in any 30-day period.
* OR History of secondary infections associated with AIDS related complex (ARC) including:
* Recurrent oral candidiasis documented by morphology or by response to antifungal therapy within 3 years.
* Herpes zoster infection within 3 years.
* Oral hairy leukoplakia at any time.
* OR History of opportunistic disease fulfilling the CDC surveillance definition of AIDS.
* Signs and symptoms at baseline characteristic of acute HIV disease (CDC group I).
* Evidence of significant neurologic dysfunction as currently defined by CDC following standard neurologic screening and AIDS Dementia Assessment.

Prior Medication:

Excluded:

- Previous treatment for greater than 3 months duration with any antiretroviral compound such as zidovudine (AZT).

Excluded within 4 weeks of study entry:

- Treatment with any potentially myelosuppressive drug, nephrotoxic agent, or other experimental therapy.

Excluded within 3 months of study entry:

- Antiretroviral drugs or biologic response modifiers.

Excluded within 4 months of study entry:

- Systemic corticosteroids.

Patients must meet the following criteria:

* HIV infection demonstrated by ELISA and confirmed by Western blot.
* Signs and symptoms of HIV disease limited to those characteristic of CDC groups II (asymptomatic) and III (persistent generalized lymphadenopathy - PGL).
* Ability to give informed consent.
* Willingness to be followed by the originating medical center for the entire 3-year duration of the study.

Active drug or alcohol abuse sufficient in the investigator's opinion to prevent compliance with the study regimen.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (22):
- United States (22):
  - LaJolla Veterans Administration Med Ctr, La Jolla, California
  - AIDS Clinical Trials Group, San Diego, California
  - Georgetown Univ Med Ctr, Washington D.C., District of Columbia
  - Univ of Miami School of Medicine, Miami, Florida
  - Univ of South Florida, Tampa, Florida
  - Emory Univ School of Medicine, Atlanta, Georgia
  - Univ of New Mexico Hlth Sciences Ctr / Dept of Med, Albuquerque, New Mexico
  - Northshore Hosp / Cornell Univ, Manhasset, New York
  - Nalle Clinic, Charlotte, North Carolina
  - Bowman Gray School of Medicine / North Carolina Baptist Hosp, Winston-Salem, North Carolina
  - Oregon Health Sciences Univ, Portland, Oregon
  - Good Samaritan Hosp, Portland, Oregon
  - Buckley Braffman Stern Med Associates, Philadelphia, Pennsylvania
  - Graduate Hosp, Philadelphia, Pennsylvania
  - Med Univ of South Carolina, Charleston, South Carolina
  - Regional Med Ctr at Memphis, Memphis, Tennessee
  - Univ TX Galveston Med Branch, Galveston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Dr Kristen Reis, Salt Lake City, Utah
  - Univ of Utah School of Medicine, Salt Lake City, Utah
  - Med College of Virginia, Richmond, Virginia
  - Milwaukee County Med Complex, Milwaukee, Wisconsin